CLINICAL TRIAL: NCT06351033
Title: Efficacy of Ozonated Oil as a Dietary Supplement in the Clinical Management of Patients With Macular Degeneration
Brief Title: Ozonized Oil as Dietary Supplement in Macular Degeneration
Status: Active, not recruiting | Type: Observational
Sponsor: Alba Di Pardo (Other)
Responsible Party: Sponsor-Investigator, Alba Di Pardo, PhD, Neuromed IRCCS
Organization: Neuromed IRCCS (Other)
Other Study IDs: ADP_012023
Record Dates: First submitted 2023-03-14; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Maculopathy
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Placebo: Placebo: control group made up of subjects affected by maculopathy - eligible according to the study protocol - subjected to traditional elective treatments only (including intravitreal Anti-VEGF injections).
- Ozonized Oil: Ozonized Oil: intervention group made up of subjects affected by maculopathy - eligible according to the study protocol - subjected to the traditional treatments of choice (including anti-VEGF intravitreal injections) who receive supplementary treatment with the intake of HOO gastro-resistant capsules.
  Interventions: Dietary Supplement: High ozonide (HOO) ozonated oil

INTERVENTIONS:
Dietary Supplement: High ozonide (HOO) ozonated oil — ozonated oil with high ozonides (HOO) administered orally (os) in gastro-resistant capsules
  Groups: Ozonized Oil

SUMMARY:
Macular degeneration, also called age-related macular degeneration (AMD), is a leading cause of visual impairment and severe vision loss.

AMD is a disease with a multifactorial etiology. The main factors which, associated with the genetic ones, increase the risk of WMD onset are represented by smoking, obesity, hypertension, cardio-vascular diseases, a diet rich in dietary fat and alcohol intake. From an organic point of view, AMD is a disease that affects the macular region of the retina, causing progressive loss of central vision.

Retinal cells are characterized by high oxygen consumption. Reactive oxygen species (ROS), such as superoxide anion, hydrogen peroxide and hydroxyl radical are the standard product of cellular metabolism within the mitochondria. Under physiological conditions, ROS are neutralized by a system of antioxidants. In case of cellular metabolism disturbances or insufficiency of the antioxidant system, an excess of ROS can be produced which contributes to oxidative stress, widely described as exerting deleterious effects on cells. The high oxygen requirement and low levels of antioxidant enzymes make the retina extremely sensitive to oxidative stress and more susceptible to cell death. Prevention of neuronal death in the retina becomes a crucial aspect for the management of WMD.

The treatment of choice for AMD today is the use of anti-VEGF (Vascular Endothelial Growth Factor) drugs, they are effective for neo-vascular AMD, acting on the inhibition of the angiogenic protein VEGF, which is produced in the retina and induced by hypoxia and other conditions. It is practice, however, to support the integration of nutritional supplements such as zinc, resveratrol, carotenoids such as lutein and zeaxanthin, vitamin E and Omega-3 fatty acids.

The aim of this study is to evaluate the efficacy of ozonated oil with high ozonides (HOO) administered orally as gastro-resistant capsules (O3Zone, GS Pharma, Malta), as an integrative and complementary treatment in patients affected by macular degeneration in the possible slowing of disease progression.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy of ozonated oil with high ozonides (HOO) administered orally as gastro-resistant capsules (O3Zone, GS Pharma, Malta), as an integrative and complementary treatment in patients affected by macular degeneration.

Field of view will be monitored to reveal the possible slowing of disease progression.

ELIGIBILITY:
Definite AMD diagnosis with documented disease progression within the past 6 months

* Age: 50-85 years old
* Ascertained differential diagnosis with the aid of diagnostic tools: fundus examination eye; analysis of the macular region using optical computed tomography (OCT)

Exclusion Criteria:

* Psychiatric diseases
* Type I and II diabetes
* Patients with high refractive defects: myopia > 6 d; hyperopia > 4 d; astigmatism > 4 d
* Corneal pathologies
* Hereditary retinal diseases
* Autoimmune diseases (uveitis)
* Glaucoma
* Oncological diseases
* Liver and kidney disease
* Inclusion in other clinical trials
* Inability to understand informed consent and the purpose of the study
* Women who are pregnant or who may become pregnant during treatment

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects participating in the study will be recruited at the Neuro-Ophthalmology Unit of the IRCCS Neuromed according to the selected inclusion and exclusion criteria. They will then be sent to genetic counseling for the reconstruction of the family genealogy, medical history collection and determination of the genetic predisposition to AMD. All recruited individuals will be entered into a database dedicated to the project.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
evaluation of any slowing down of the maculopathy | 3 months from the beginning of the ozonated oil administration
  field of view
evaluation of any slowing down of the maculopathy | 6 months from the beginning of the ozonated oil administration
  field of view
evaluation of any slowing down of the maculopathy | 9 months from the beginning of the ozonated oil administration
  field of view
evaluation of any slowing down of the maculopathy and closure of the study | 12 months from the beginning of the ozonated oil administration
  field of view

CONTACTS AND LOCATIONS:
Overall Officials: Eliana Palermo, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Italy